CLINICAL TRIAL: NCT03454698
Title: A Targeted Interprofessional Education Intervention to Address Therapeutic Adherence of Venous Leg Ulcer Persons (TIEIVLU): Study Protocol for a Randomized Controlled Trail
Brief Title: Education for Venous Leg Ulcer Patients
Acronym: legulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: School of Health Sciences Geneva (Other)
Responsible Party: Principal Investigator, Sebastian Probst, Clinical Professor, School of Health Sciences Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: leg_ulcer_intervention
Record Dates: First submitted 2018-02-07; First posted 2018-03-06 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Interprofessional Education for Venous Leg Ulcer Patients
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contol (Other): "Usual care" for patients in the CG is defined as follows: Visits to the outpatient wound-care centre as directed by a physician. Wound care performed by the wound expert according to the hospital's own standards. This standard corresponds to the one from the EWMA.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — "Usual care" as described for the CG also applies to the IG. The intervention will consist of giving patients an opportunity to learn about the use of compression bandages, wearing and putting on compression stockings, physical activity, good skin care, and a high-protein, vitamin-rich diet. This group will be supervised by a study nurse, who will not be identical with the nurse in charge of the control group.

SUMMARY:
Venous leg ulcers (VLU) are slow healing wounds. They have a high recurrence rate and are associated with pain, infection, smell and exudate. 60% of VLU become chronic. Current therapeutic approaches are multifaceted and focus on improving wound healing and preventing recurrences. As those approaches include compression therapy, leg elevation, specific exercises for the foot/ ankle region and a protein rich diet/ nutrition plan a multidisciplinary team of health care professionals such as nursing, physiotherapy, occupational therapy and nutrition specialists. Most persons with VLU have a knowledge deficit in regards to therapeutic measures and hence have difficulties with adherence to treatment protocols/ management plans. It is of utmost importance, and best practice, that the treatment team provides effective patient education and support during the learning phase.

However, there is little evidence and no published studies that describe and evaluate effective multidisciplinary educational interventions that target compliance/ adherence to the treatment plan in patients with VLU. Therefore the investigators propose to develop an evidence-based interprofessional educational intervention and evaluate its feasibility first in a pilot study and subsequently in a randomized controlled trail.

Method/Design: Firstly, the development of an evidence based education intervention in collaboration with an expert panel and secondly a randomized controlled pilot study in one wound care outpatient clinic is proposed. Data will be analyzed using SPSS version 23. Univariate and bivariate analysis will be conducted according to the data level and distribution of the data.

Discussion: The TIEIVLU will firstly develop an evidenced based educational intervention and secondly examine the feasibility of implementing this education intervention in a realistic care context in patients with VLU. The results will inform the final design of a following RCT which will examine the effectiveness of the educational intervention. An intervention that enhances patient adherence to therapy and hence reduces the negative outcomes of VLU would be beneficial to individual patients as well as society as a whole.

DETAILED DESCRIPTION:
Background: Venous leg ulcers (VLU) are slow healing wounds. They have a high recurrence rate and are associated with pain, infection, smell and exudate. 60% of VLU become chronic. The signs and symptoms of VLU are not only a burden on those who are affected by it but also on the health care system and society in general. While the prevalence of VLU in the general population is 1%, it rises to 3% in the over 80 age group. The cost of treatment and care for VLU is estimated to be 2 to 3% of the overall health expenditure. Current therapeutic approaches are multifaceted and focus on improving wound healing and preventing recurrences. As those approaches include compression therapy, leg elevation, specific exercises for the foot/ ankle region and a protein rich diet/ nutrition plan a multidisciplinary team of health care professionals such as nursing, physiotherapy, occupational therapy and nutrition specialists. Most person with VLU have a knowledge deficit in regards to therapeutic measures and hence have difficulties with adherence to treatment protocols/ management plans. It is of utmost importance, and best practice, that the treatment team provides effective patient education and support during the learning phase.

However, there is little evidence and no published studies that describe and evaluate effective multidisciplinary educational interventions that target compliance/ adherence to the treatment plan in patients with VLU. Therefore the investigators propose to develop an evidence-based interprofessional educational intervention and evaluate its feasibility first in a pilot study and subsequently in a randomized controlled trail.

Method/Design: Firstly, the development of an evidence based education intervention in collaboration with an expert panel and secondly a randomized controlled pilot study in one wound care outpatient clinic is proposed. Data will be analyzed using SPSS version 23. Univariate and bivariate analysis will be conducted according to the data level and distribution of the data.

Discussion: The TIEIVLU will firstly develop an evidenced based educational intervention and secondly examine the feasibility of implementing this education intervention in a realistic care context in patients with VLU. The results will inform the final design of a following RCT which will examine the effectiveness of the educational intervention. An intervention that enhances patient adherence to therapy and hence reduces the negative outcomes of VLU would be beneficial to individual patients as well as society as a whole.

ELIGIBILITY:
Inclusion Criteria:

* An existing open venous leg ulcer
* An ankle brachial pressure index (ABPI) between 0.8 and 1.3
* Age over 18 years
* Proficiency in the French language

Exclusion Criteria:

* Valid informed consent is not or cannot be given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
acceptability of an interprofessional education for venous leg ulcer patients | 3 months
  acceptability of this elaborated interprofessional education

CONTACTS AND LOCATIONS:
Locations (1):
- Cité Génération Maison de santé, Onex, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Probst S, Allet L, Depeyre J, Colin S, Buehrer Skinner M. A targeted interprofessional educational intervention to address therapeutic adherence of venous leg ulcer persons (TIEIVLU): study protocol for a randomized controlled trial. Trials. 2019 Apr 29;20(1):243. doi: 10.1186/s13063-019-3333-4. PMID 31036037